CLINICAL TRIAL: NCT06612801
Title: REThinkGame4training: Training Emotion Regulation Abilities Using an Online Therapeutic Game
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Responsible Party: Principal Investigator, Oana David, Professor Ph.D, Babes-Bolyai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REThinkGame4training
Record Dates: First submitted 2024-09-23; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Emotion Regulation Abilities
Keywords: online game; therapeutic game; digital intervention; REThink game; emotion regulation abilities; irrationality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: REThink therapeutic game (Experimental): Participants in the experimental group will received the game-based intervention called REThink Game
  Interventions: Behavioral: The REThink Game
- Control: Care as usual (No Intervention): Participants in the control group do not receive an intervention but they have access to standard resources from the school

INTERVENTIONS:
Behavioral: The REThink Game — REThink is an online therapeutic game designed to improve the emotional well-being of young people, based on the principles of Rational Emotive Behavior Therapy (REBT). The game features a character named RETMAN, who leads players through seven levels, each dedicated to teaching a particular emotional regulation skill. Each level consists of three sub-levels that gradually become more challenging. REThink can be utilized as a standalone intervention, as a complement to self-help psychotherapeutic methods, or for focused skills training in emotional regulation. Each level trains a specific emoion-regulation skills such as emotion recognition, relaxation, cognitive change, problem solving, compassion and self-compassion.
  Arms: Experimental: REThink therapeutic game

SUMMARY:
To test the efficacy of the REThink therapeutic game in training emotion regulation abilities of children and adolescents.

DETAILED DESCRIPTION:
The primary aim of this study is to evaluate the effectiveness of the REThink therapeutic game in training emotion regulation abilities in children aged 8 to 12 years. The participants will be recruitedfrom various schools and counties, ensuring a diverse sample. Those in the experimental group will engage with the REThink game over a four-week period. To assess the impact of the intervention, standardized pre-test and post-test measures will be administered, allowing for a comparison of mental health outcomes before and after the use of the therapeutic game. The study seeks to determine whether this digital tool can serve as an effective training for improving emotion regulation abilities in this age group.

ELIGIBILITY:
Inclusion Criteria:

* children and adolescents aged 8 to 12 years
* non-clinical levels of mental health symptoms on any SDQ subscale or total score
* parental consent provided

Exclusion Criteria:

* intellectual disability or physical limitations precluding the use of the online game
* does not have parental informed consent
* clinical or subclinical level on the SDQ measure, total score, or any subscale

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 237 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Emotion regulation abilities | baseline assessment, one week before starting the intervention
  The Emotion Regulation Index for Children and Adolescents (ERICA; Biesecker & Easterbrooks, 2001). The 13 items are measured on a five-point Likert scale, from 0 -strong disagreement to 5 - strong agreement-; where higher scores represent better emotional regulation abilities. The scale has two subscales namely, emotional control ( lowest score 8 and highest 40) and emotional awareness subscales (lowest score 5, and highest 25).
Changes in emotion regulation abilities | post-test assessment, one week after finishing the intervention
  The Emotion Regulation Index for Children and Adolescents (ERICA; Biesecker &amp; Easterbrooks, 2001). The 13 items are measured on a five-point Likert scale, from 0 -strong disagreement to 5 - strong agreement-; where higher scores represent better emotional regulation abilities. The scale has two subscales namely, emotional control ( lowest score 8 and highest 40) and emotional awareness subscales (lowest score 5, and highest 25).
Irrationality | baseline assessment, one week before starting the intervention
  The Child and Adolescent Scale of Irrationality (CASI, Bernard & Cronan, 1999) will be used in order to test irrational/rational beliefs as a mechanism of change. Children and adolescents were asked to express their agreement/disagreement with the 28 statements on a 5-point Likert-type scale, from 1 ("strong disagreement") to 5 ("strong agreement"). The minimum score is 28 and the maximum score is 140. Higher scores represent higher levels of irrationality.
Changes in irrationality | post-test assessment, one week after finishing the intervention
  The Child and Adolescent Scale of Irrationality (CASI, Bernard & Cronan, 1999) will be used in order to test irrational/rational beliefs as a mechanism of change. Children and adolescents were asked to express their agreement/disagreement with the 28 statements on a 5-point Likert-type scale, from 1 ("strong disagreement") to 5 ("strong agreement"). The minimum score is 28 and the maximum score is 140. Higher scores represent higher levels of irrationality.

OTHER OUTCOMES:
Mental health symthoms | baseline assessment, inclusion criteria
  Strengths and Difficulties Questionnaire (SDQ; Goodman, 1997). The scale has 25-items within its five subscales, namely emotional symptoms (ES), conduct problems (CP), hyperactivity/inattention (HY), peer relationship (PR) problems and prosocial behavior (PS) and total mental health difficulties score (MHD). The items are rated on a 3-point Likert scale, from 0 (not true) to 2 (certainly true). The minimum score is 0 and the maximum is 40. Higher scores represent higher level of mental health difficulties.

CONTACTS AND LOCATIONS:
Locations (1):
- Babes-Bolyai University, Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: No